CLINICAL TRIAL: NCT05195671
Title: Implications of Ethics Determinant on Dentistry and Pharmacy Research: A Study of IRB Perspective
Brief Title: Implications of Ethics Determinant on Dentistry and Pharmacy Research
Status: Completed | Type: Observational
Sponsor: Misr International University (Other)
Responsible Party: Sponsor
Other Study IDs: ETH12
Record Dates: First submitted 2021-12-27; First posted 2022-01-19 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2021-12

CONDITIONS: Review, Research Peer
Keywords: Dental Ethics; Pharmacy Ethics; Institutional Ethics Committees

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Review — Reviewing all protocols

SUMMARY:
The ethical review of dental and pharmacy research protocols has its own challenges facing the institutional ethical committees. Seemingly low risk procedure might pose controversies among committees' members. The aim of this article is to describe some of the ethical concerns, particular to dental and pharmacy research that an ethics committee could face while reviewing dental research.

DETAILED DESCRIPTION:
The investigators have read all protocols submitted to the MIU IRB and reviewed all meetings' minutes to outline the ethical concerns that warranted discussions in the meetings, and how the committee came to a resolution for those concerns.

ELIGIBILITY:
Inclusion Criteria:

* all protocols submitted to IRB

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All students' research, Post-Grad and Research protocols submitted to MIU Institutional Review Board
Sampling Method: Non-Probability Sample
Enrollment: 131 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-10 (Actual)

PRIMARY OUTCOMES:
Ethical concerns | 1 month
  Frequencies and percentages of ethical concerns

CONTACTS AND LOCATIONS:
Overall Officials: Mahassen M Farghaly, Professor, Study Director — Vice president of community services and environmental awareness
Locations (1):
- Misr International University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] 1- Allison M. DiMatteo, BA, MP. The Legacy of Dental Research. Inside Dentistry. 2006, June; (2), Issue 5.
- [Background] Gillett GR. Ethics and dental research. J Dent Res. 1994 Nov;73(11):1766-72. doi: 10.1177/00220345940730111401. PMID 7983264
- [Background] Navabi N, Shahravan A, Modaberi A. Reporting of Ethical Considerations Associated with Clinical Trials Published in Iranian Dental Journals between 2001 and 2011. Iran J Public Health. 2013 Jun 1;42(6):594-601. eCollection 2013. PMID 23967427
- [Background] Mancl LA, Leroux BG, DeRouen TA. Between-subject and within-subject statistical information in dental research. J Dent Res. 2000 Oct;79(10):1778-81. doi: 10.1177/00220345000790100801. PMID 11077994
- [Background] Burt BA. Concepts of risk in dental public health. Community Dent Oral Epidemiol. 2005 Aug;33(4):240-7. doi: 10.1111/j.1600-0528.2005.00231.x. PMID 16008630
- [Background] Naik SP, Nividan KS, Pinto B, Shobha R, Dutt AS, and Rahul N. Ethical Issue and Challenges in Dentistry. International Journal of Preventive and Clinical Dental Research. 2016 October - December; 3(4): 285-87
- [Background] El-Dessouky HF, Abdel-Aziz AM, Ibrahim C, Moni M, Abul Fadl R, Silverman H. Knowledge, Awareness, and Attitudes about Research Ethics among Dental Faculty in the Middle East: A Pilot Study. Int J Dent. 2011;2011:694759. doi: 10.1155/2011/694759. Epub 2011 Jul 3. PMID 21754933
- [Background] Deolia SG, Prasad K, Chhabra KG, Kalyanpur R, Kalghatgi S. An Insight Into Research Ethics among Dental Professionals in A Dental Institute, India- A Pilot Study. J Clin Diagn Res. 2014 Sep;8(9):ZC11-4. doi: 10.7860/JCDR/2014/10118.4794. Epub 2014 Sep 20. PMID 25386512
- [Background] Dube-Baril C. The personalized consent form: an optional, but useful tool! J Can Dent Assoc. 2004 Feb;70(2):89-92. PMID 14756938
- [Background] Fitzgerald DW, Marotte C, Verdier RI, Johnson WD Jr, Pape JW. Comprehension during informed consent in a less-developed country. Lancet. 2002 Oct 26;360(9342):1301-2. doi: 10.1016/S0140-6736(02)11338-9. PMID 12414207
- [Background] Kadam RA. Informed consent process: A step further towards making it meaningful! Perspect Clin Res. 2017 Jul-Sep;8(3):107-112. doi: 10.4103/picr.PICR_147_16. PMID 28828304
- [Background] Khallof RO, Doumani M, Farid FAS, Mostafa D, Alhafian RAA. Dental education in the Arabic language vs English language: A survey among Arab dentists. J Family Med Prim Care. 2019 Dec 10;8(12):3908-3914. doi: 10.4103/jfmpc.jfmpc_572_19. eCollection 2019 Dec. PMID 31879634
- [Background] Hon YK, Narayanan P, Goh PP. Extended discussion of information for informed consent for participation in clinical trials. The Cochrane Database of Systematic Reviews. 2017 (8).
- [Background] Lasers in Dentistry: A Review Chaya M David1, Pankaj Gupta; International Journal of Advanced Health Sciences • Vol 2 Issue 8 • December 2015, 7-13
- See also: Principles of patient consent. London: 2009. General Dental Council — http://www.gdc-uk.org
- See also: Ethnologue: languages of the world. Texas: 2021. SIL International. — http://www.ethnologue.com